CLINICAL TRIAL: NCT01860573
Title: Neurodevelopmental and Growth Outcomes of Early, Aggressive Protein Intake in Very Low Birthweight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Joseph Bliss, Staff Neonatologist, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0089
Record Dates: First submitted 2013-05-14; First posted 2013-05-22 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Prematurity
Keywords: Amino acids; Protein
MeSH Terms: conditions — Premature Birth | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard amino acids (Active Comparator): Receive 1-2 gm/kg/day amino acids at birth and advanced by 0.5 gm/kg/day for goal of 4 gm/kg/day
  Interventions: Drug: Amino acids
- High amino acids (Experimental): Receive 3-4 gm/kg/day amino acids at birth and advanced to goal of 4 gm/kg/day as soon as possible after birth
  Interventions: Drug: Amino acids

INTERVENTIONS:
Drug: Amino acids
  Other Names: Premasol

SUMMARY:
The purpose of this study is to determine whether providing increased protein to premature infants in the first week of life allows for better growth during the hospital stay and improved developmental outcomes by age 2.

ELIGIBILITY:
Inclusion Criteria:

* birth weight 400 to 1250 grams
* 24 0/7 to 30 6/7 weeks gestational age

Exclusion Criteria:

* chromosomal, structural, metabolic, endocrine, or renal abnormalities that could affect growth
* infants >18 hours of age
* infants in extremis who are unlikely to survive past 72 hours

Max Age: 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-11; Primary Completion 2013-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Bliss, MD, PhD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Poindexter BB, Langer JC, Dusick AM, Ehrenkranz RA; National Institute of Child Health and Human Development Neonatal Research Network. Early provision of parenteral amino acids in extremely low birth weight infants: relation to growth and neurodevelopmental outcome. J Pediatr. 2006 Mar;148(3):300-305. doi: 10.1016/j.jpeds.2005.10.038. PMID 16615955
- [Background] Stephens BE, Walden RV, Gargus RA, Tucker R, McKinley L, Mance M, Nye J, Vohr BR. First-week protein and energy intakes are associated with 18-month developmental outcomes in extremely low birth weight infants. Pediatrics. 2009 May;123(5):1337-43. doi: 10.1542/peds.2008-0211. PMID 19403500
- [Background] Thureen PJ, Melara D, Fennessey PV, Hay WW Jr. Effect of low versus high intravenous amino acid intake on very low birth weight infants in the early neonatal period. Pediatr Res. 2003 Jan;53(1):24-32. doi: 10.1203/00006450-200301000-00008. PMID 12508078
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Amino Acids: Receive 1-2 gm/kg/day amino acids at birth and advanced by 0.5 gm/kg/day for goal of 4 gm/kg/day
  Amino acids
- High Amino Acids: Receive 3-4 gm/kg/day amino acids at birth and advanced to goal of 4 gm/kg/day as soon as possible after birth
  Amino acids
Period: Overall Study
Arm/Group | Standard Amino Acids | High Amino Acids
Started | 83 | 85
Completed | 83 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Amino Acids | High Amino Acids | Total
Number analyzed (Participants) | 83 | 85 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 83 | 85 | 168
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 46 | 83
  Male | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Weight<10th Percentile for Age
Time Frame: 36 weeks post-conceptual age
Population: Data not available for subjects who died or were discharged prior to 36 weeks post-conceptual age
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 67 | 72
Participants | 32 | 41

2. Primary Outcome: Number of Participants With Length <10th Percentile for Age
Time Frame: 36 weeks post-conceptual age
Population: Data not available for subjects who died or were discharged prior to 36 weeks post-conceptual age, and some data were missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 60 | 63
Participants | 29 | 42

3. Primary Outcome: Number of Participants With Head Circumference <10th Percentile for Age
Time Frame: 36 weeks post-conceptual age
Population: Data not available for subjects who died or were discharged prior to 36 weeks post-conceptual age and some data were missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 67 | 68
Participants | 20 | 23

4. Primary Outcome: Cognitive Development Score
Description: Reported as units on a scale with mean of 100 and a Standard Deviation of 15, and range from 40-160. Higher values indicate a better outcome.
Time Frame: 18-22 months corrected gestational age
Population: Data not available for subjects who died or were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 59 | 55
units on a scale | 90.2 (10.3) | 90.6 (12.7)

5. Secondary Outcome: Serum Bicarbonate
Time Frame: Day of life 1, 2, 3, 5 and 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 83 | 85
mmol/L
  Day 1 | 21.2 (2.9) | 21.8 (2.4)
  Day 2 | 20.7 (3.1) | 21.2 (3.2)
  Day 3 | 20.0 (3.5) | 20.1 (3.7)
  Day 5 | 18.7 (4.0) | 18.0 (4.1)
  Day 7 | 18.7 (4.0) | 18.3 (4.4)

6. Secondary Outcome: Serum Creatinine
Time Frame: Day of life 1, 2, 3, 5 and 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 83 | 85
mg/dL
  Day 1 | .99 (.20) | .97 (.19)
  Day 2 | 1.11 (.22) | 1.11 (.28)
  Day 3 | 1.16 (.26) | 1.10 (.28)
  Day 5 | 1.18 (.26) | 1.07 (.31)
  Day 7 | 1.01 (.27) | .93 (.27)

7. Secondary Outcome: Serum Blood Urea Nitrogen
Time Frame: Day of life 1, 2, 3, 5 and 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Amino Acids | High Amino Acids
Number analyzed (Participants) | 83 | 85
mg/dL
  Day 1 | 19.0 (7.2) | 21.6 (8.0)
  Day 2 | 26.1 (8.8) | 35.8 (9.7)
  Day 3 | 29.8 (10.6) | 43.9 (14.3)
  Day 5 | 35.3 (15.5) | 49.1 (17.5)
  Day 7 | 32.9 (15.9) | 38.9 (19.3)

ADVERSE EVENTS:
Description: Participants who died were not able to be assessed for the other (not including serious) adverse events reported, because these adverse events are captured later in hospitalization. Thus, the total infants at risk for other adverse events is fewer than the number at risk for serious adverse events.
Arm/Group | Standard Amino Acids | High Amino Acids
Serious Adverse Events (participants affected / at risk) | 31/83 | 19/85
Other Adverse Events (participants affected / at risk) | 35/73 | 32/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Amino Acids (N=83) | High Amino Acids (N=85)
Death (Pregnancy, puerperium and perinatal conditions) | 10 | 9
Sepsis (Infections and infestations) | 31 | 19
Necrotizing Enterocolitis (Gastrointestinal disorders) | 15 | 13
Intaventricular Hemorrhage Grade III/IV (Nervous system disorders) | 7 | 4
Periventricular Leukomalacia (Nervous system disorders) | 5 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Amino Acids (N=73) | High Amino Acids (N=74)
Retinopathy of Prematurity (Eye disorders) | 35 | 29
Bronchopulmonary Dysplasia (Respiratory, thoracic and mediastinal disorders) | 32 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes